CLINICAL TRIAL: NCT01431092
Title: Prolonged-release Melatonin Versus Placebo for Benzodiazepine Discontinuation in Patients With Schizophrenia: a Randomized Clinical Trial
Brief Title: Melatonin Versus Placebo for Benzodiazepine Discontinuation in Patients With Schizophrenia
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lone Baandrup (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Lone Baandrup, MD, Ph.D., University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-024065-46; 2010-024065-46 (EudraCT Number)
Record Dates: First submitted 2011-08-31; First posted 2011-09-09 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Both Circadin and placebo are encapsulated in lactose containing gelatin capsules to optimize the blinding.
  Arms: Placebo
Drug: Melatonin — Prolonged-release melatonin (Circadin®) 2 mg, once daily, 1-2 hours before bedtime.
  Other Names: Prolonged-release melatonin; Circadin®
  Arms: Melatonin

SUMMARY:
In this trial, researchers aim to investigate if prolonged-release melatonin can facilitate the withdrawal of chronic benzodiazepine administration in patients with schizophrenia. Furthermore, researchers will investigate the association of benzodiazepine dose reduction with the following clinically important variables: sleep, psychophysiology, cognition, social function, and quality of life.

DETAILED DESCRIPTION:
Treatment of schizophrenia frequently includes prolonged administration of benzodiazepines despite lack of evidence of its use. It is often difficult to discontinue use of benzodiazepines because of development of dependence.

After being randomized to prolonged-release melatonin (Circadin®) 2 mg daily versus matching placebo, participants are required to slowly taper off their benzodiazepine dose towards no intake. Data are collected at baseline and at 6 months follow-up regarding medical treatment, cognition, psychophysiology, sleep, laboratory tests, adverse events, psychopathology, social function, and quality of life. Data on medical treatment, cognition, adverse events, social function, and quality of life are also collected at 2 and 4 months follow-up.

The results from this trial will assess if melatonin has a role in withdrawing long-term benzodiazepine administration in schizophrenia patients. This group of patients is difficult to treat and therefore often subject to polypharmacy which may play a role in the reduced life expectancy compared to the background population. In addition, the data of the trial are also analyzed as an observational cohort design to investigate the association of benzodiazepine dose reduction/discontinuation with psychophysiology, cognition, sleep, quality of life, and other selected variables (not further described below, see trial protocol). Knowledge of these important clinical aspects is lacking in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia, schizoaffective disorder, or bipolar affective disorder (ICD-10 criteria for schizophrenia (F20), schizoaffective disorder (F25) or bipolar affective disorder (F31) must be fulfilled at inclusion or previously as documented by chart review; fulfillment of relevant DSM-IV-TR criteria will also be registered).
* Treated with the same antipsychotic drug for at least 3 months before inclusion (change of dose, antipsychotic polypharmacy and prescription/discontinuation of add-on drugs allowed but the basic antipsychotic treatment should be the same).
* Continuously treated with at least one benzodiazepine (chlordiazepoxide, diazepam, clobazam, clonazepam, flunitrazepam, nitrazepam, bromazepam, alprazolam, lorazepam, lormetazepam, oxazepam, triazolam) or benzodiazepine related drug (zolpidem, zopiclone, zaleplon) for at least 3 months before inclusion.
* Age 18+.
* Fertile women: negative pregnancy test at baseline and use of safe contraceptives (intrauterine devices or hormonal contraception) throughout the trial period and 1 day after withdrawal of trial medication. This does not apply to sterile or infertile participants, i.e. surgically sterilized or post menopausal (missing period for at least 12 months before inclusion) women.
* Written informed consent.

Exclusion Criteria:

* Known aggressive or violent behavior.
* Mental retardation, pervasive developmental disorder, or dementia.
* Epilepsy, terminal illness, severe comorbidity or unable to understand Danish.
* Allergic to compounds in the trial medication (melatonin, lactose, starch, gelatin, talc).
* Hepatic impairment (known diagnosis).
* Pregnancy and nursing.
* Missing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Benzodiazepine (including benzodiazepine related drugs) dose at 6 months follow-up. | 6 months follow-up.
  The general linear model is used with the outcome measure (dose after 6 months) as the dependent variable and the indicator of intervention and the baseline value as the independent variables. If the assumptions of the model cannot be fulfilled either directly or after transformation a non-parametric method will be used.

SECONDARY OUTCOMES:
Pattern of benzodiazepine dose over time. | 2, 4, and 6 months.
  The mixed model with repeated measures will be used to analyze the time course. The model is outcome measure = int + baseline + a*t + b*t*t + c*baseline*t + d*baseline*t*t + e*I + f*I*t + g*I*t*t where t is time, I the intervention indicator, int the intercept, and a through g the coefficients. Using Akaike's criterium the best co-variance matrix is first chosen among an unstructured, a compound symmetric, or a first order autoregressive.
The fraction of participants who has completely discontinued benzodiazepines 6 months after initiating trial medication. | 6 months follow-up.
  The analysis will be done using a logistic regression model where logit(p) is the dependent variable, p is the probability of completing the withdrawal, and a binary intervention indicator is the independent variable.
Pattern of P300 amplitude (psychophysiology) over time. | 2, 4, and 6 months.
  The mixed model with repeated measures will be used to analyze the time course. The model is outcome measure = int + baseline + a*t + b*t*t + c*baseline*t + d*baseline*t*t + e*I + f*I*t + g*I*t*t where t is time, I the intervention indicator, int the intercept, and a through g the coefficients. Using Akaike's criterium the best co-variance matrix is first chosen among an unstructured, a compound symmetric, or a first order autoregressive.
Pattern of Brief Assessment of Cognition in Schizophrenia (BACS) composite score over time. | 2, 4, and 6 months.
  The mixed model with repeated measures will be used to analyze the time course. The model is outcome measure = int + baseline + a*t + b*t*t + c*baseline*t + d*baseline*t*t + e*I + f*I*t + g*I*t*t where t is time, I the intervention indicator, int the intercept, and a through g the coefficients. Using Akaike's criterium the best co-variance matrix is first chosen among an unstructured, a compound symmetric, or a first order autoregressive.
Sleep efficiency (polysomnography) at 6 months follow-up. | 6 months.
  The general linear model is used with the outcome measure (sleep efficiency) as the dependent variable and the indicator of intervention and the baseline value as the independent variables. If the assumptions of the model cannot be fulfilled either directly or after transformation a non-parametric method will be used.
Pittsburgh Sleep Quality Index (PSQI) global score at 6 months follow-up. | 6 months.
  The general linear model is used with the outcome measure (PSQI) as the dependent variable and the indicator of intervention and the baseline value as the independent variables. If the assumptions of the model cannot be fulfilled either directly or after transformation a non-parametric method will be used.
Pattern of Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ-2) score over time. | 2, 4, and 6 months.
  The mixed model with repeated measures will be used to analyze the time course. The model is outcome measure = int + baseline + a*t + b*t*t + c*baseline*t + d*baseline*t*t + e*I + f*I*t + g*I*t*t where t is time, I the intervention indicator, int the intercept, and a through g the coefficients. Using Akaike's criterium the best co-variance matrix is first chosen among an unstructured, a compound symmetric or a first order autoregressive.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Baandrup, MD, PhD, Principal Investigator — CNSR/CINS; Birte Glenthøj, MD, MSc, Study Chair — CNSR/CINS
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research (CNSR)/Center for Clinical Intervention and Neuropsychiatric Schizophrenia Research (CINS), University of Copenhagen, Mental Health Centre Glostrup, Mental Health Services - Capital Region of Denmark, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Volz A, Khorsand V, Gillies D, Leucht S. Benzodiazepines for schizophrenia. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD006391. doi: 10.1002/14651858.CD006391. PMID 17253592
- [Background] Monti JM, Monti D. Sleep disturbance in schizophrenia. Int Rev Psychiatry. 2005 Aug;17(4):247-53. doi: 10.1080/09540260500104516. PMID 16194796
- [Background] Buscemi N, Vandermeer B, Hooton N, Pandya R, Tjosvold L, Hartling L, Vohra S, Klassen TP, Baker G. Efficacy and safety of exogenous melatonin for secondary sleep disorders and sleep disorders accompanying sleep restriction: meta-analysis. BMJ. 2006 Feb 18;332(7538):385-93. doi: 10.1136/bmj.38731.532766.F6. Epub 2006 Feb 10. PMID 16473858
- [Background] Shamir E, Laudon M, Barak Y, Anis Y, Rotenberg V, Elizur A, Zisapel N. Melatonin improves sleep quality of patients with chronic schizophrenia. J Clin Psychiatry. 2000 May;61(5):373-7. doi: 10.4088/jcp.v61n0509. PMID 10847313
- [Background] Suresh Kumar PN, Andrade C, Bhakta SG, Singh NM. Melatonin in schizophrenic outpatients with insomnia: a double-blind, placebo-controlled study. J Clin Psychiatry. 2007 Feb;68(2):237-41. doi: 10.4088/jcp.v68n0208. PMID 17335321
- [Background] Garfinkel D, Zisapel N, Wainstein J, Laudon M. Facilitation of benzodiazepine discontinuation by melatonin: a new clinical approach. Arch Intern Med. 1999 Nov 8;159(20):2456-60. doi: 10.1001/archinte.159.20.2456. PMID 10665894
- [Derived] Baandrup L, Fasmer OB, Glenthoj BY, Jennum PJ. Circadian rest-activity rhythms during benzodiazepine tapering covered by melatonin versus placebo add-on: data derived from a randomized clinical trial. BMC Psychiatry. 2016 Oct 13;16(1):348. doi: 10.1186/s12888-016-1062-8. PMID 27737649
- [Derived] Baandrup L, Fagerlund B, Jennum P, Lublin H, Hansen JL, Winkel P, Gluud C, Oranje B, Glenthoj BY. Prolonged-release melatonin versus placebo for benzodiazepine discontinuation in patients with schizophrenia: a randomized clinical trial - the SMART trial protocol. BMC Psychiatry. 2011 Oct 5;11:160. doi: 10.1186/1471-244X-11-160. PMID 21975110